CLINICAL TRIAL: NCT03304223
Title: A Proof of Concept Study for [18F]FB-IL2 PET Imaging of Infiltrating T Cells After Renal Transplantation; a Diagnostic Tool for Acute Rejection
Brief Title: IL2 Imaging in Renal Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, J.S.F. Sanders, MD, PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201501004
Record Dates: First submitted 2017-09-22; First posted 2017-10-06 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]FB-IL2 PET scan (Experimental): Renal transplant recipients with a clinical suspicion for renal transplant rejection.
  Interventions: Diagnostic Test: [18F]FB-IL2 PET scan

INTERVENTIONS:
Diagnostic Test: [18F]FB-IL2 PET scan — [18F]FB-IL2 PET scan procedure

SUMMARY:
After renal transplantation 5 to 10% of patients experience allograft rejection. Rapid and accurate diagnosis is vital for implementation of additional immunosuppressive therapy. Currently, a renal biopsy is essential for the diagnosis of renal allograft rejection. However, this is an intervention associated with complications like bleeding, patient discomfort and hospital admission. Additionally, limited biopsy sample size may lead to false negative results. So, the introduction of a new non-invasive diagnostic tool for allograft rejection could have major implications for the care of renal transplant recipients. For the purpose of visualizing infiltrating T lymphocytes with positron emission tomography (PET), the tracer 18-Fluor-Interleukin-2 ([18F]FB-IL2) has been developed. The investigators hypothesized that a high correlation exists between [18F]FB-IL2 uptake and the extend of T cell infiltration into renal transplants with signs of rejection

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged between 18 and 80 years.
* Renal Transplant recipients
* The patient understands the purpose and risks of the study and has given written informed consent to participate in the study.
* All patients will have a clinical indication for renal biopsy.

Exclusion Criteria:

* Patients with multiple-organ transplants.
* Female patients who are pregnant or unwilling to use adequate contraception during the study.
* Claustrophobia
* Altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* A clinical reason for an immediate start of a therapeutic intervention with immunosuppressive medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The ability of the [18F]FB-IL2 PET to detect renal transplant rejection | At study day 2, when PET procedure is performed.
  Uptake of [18F]FB-IL2 in the renal transplant will be correlated to inflammatory infiltrate and histological BANFF score.

SECONDARY OUTCOMES:
Uptake of [18F]FB-IL2 and correlation with renal function | At study day 2, when PET procedure is performed.
  Uptake of [18F]FB-IL2 in the renal transplant will be correlated to renal function as measured by 24-hours urine clearance and the Modification of Diet in Renal Disease equation (MDRD).
Uptake of [18F]FB-IL2 and correlation with T-cell subpopulations | At study day 2, when PET procedure is performed.
  Uptake of [18F]FB-IL2 in the renal transplant will be correlated to T-cell subpopulations in urine and blood.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Stephan F Sanders, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided